CLINICAL TRIAL: NCT04057690
Title: Automatic Prediction of Malignant Brain Edema After Middle Cerebral Artery Ischemic -Stroke
Brief Title: Automatic PredICtion of Edema After Stroke
Acronym: APICES
Status: Active, not recruiting | Type: Observational
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Other Study IDs: APICES
Record Dates: First submitted 2019-04-25; First posted 2019-08-15 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Stroke, Acute; Brain Edema
Keywords: Malignant Brain Edema; Stroke, Acute; Prediction
MeSH Terms: conditions — Stroke; Brain Edema

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- MCA ischemia without malignant edema: MCA ischemia without malignant edema
- MCA ischemia with malignant edema: MCA ischemia without malignant edema w/o surgical treatment

SUMMARY:
To use machine learning for early detection of malignant brain edema in patients with MCA ischemia

DETAILED DESCRIPTION:
Malignant cerebral edema following large ischemic strokes account for up to 10% of all ischemic strokes. Mortality rates are high and most of the survivors are left severely disabled. Although decompressive craniectomy has been shown to significantly decrease mortality, high morbidity rates among survivors are reported. The optimal timepoint when neurosurgical decompression should be performed in the individual patient varies and is a subject of debate.

Early prediction of malignant brain edema to identify those patients who benefit from surgical treatment is a clinical challenge. The aim of this study is to use machine learning for comprehensive analysis of CT images as well as clinical data from 1500 patients with large ischemic MCA strokes in oder to develop a model for early prediction of malignant brain edema. In a first step algorithms automatically identify characteristic imaging features and clinical data of 1400 retrospective data sets to create a multistage model (learning phase). This is followed by a validation phase where the model is tested with 100 other retrospective data sets.

ELIGIBILITY:
Inclusion Criteria:

* Acute ≥ subtotal MCA infarct (M1-M2 occlusion)
* with or without malignant brain swelling
* with or without reperfusion therapy
* with or without neurosurgical decompression
* with or without death following malignant brain edema

Exclusion Criteria:

* Non-acute MCA infarct
* < subtotal MCA infarct

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 1500 retrospective datasets will be collected from 5 large German stroke units. Data sets include imaging data and clinical data from patients with subtotal MCA infarcts (M1-M2 occlusion), with or without malignant brain swelling, with or without reperfusion therapy, with or without neurosurgical decompression, and with or without death following malignant brain edema. Data sets from patients who have died following malignant brain edema will be included. Each data set consists of initial NCCT, CTA, (DSA if available), and follow-up NCCT until 14 days after stroke onset as well as clinical data.
Sampling Method: Non-Probability Sample
Enrollment: 1687 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of patients with stroke-related malignant edema after recanalization treatment detected by deep learning algorithms | 4/2019-3/2022
  Deep learning algorithms will be used for automatic identification of specific image findings and specific clinical data that indicate a stroke-related malignant edema. Primary outcome measures are Sensitivity/Specificity/negative predictive value/positive predictive value of early detection of patients developing stroke-related malignant edema based on initial CT and 24 hour follow up CT and clinical parameters.

SECONDARY OUTCOMES:
Number of correctly identified specific imaging findings for early detection of malignant edema | 4/2019-3/2022
  Used specific imaging findings for early detection of malignant brain edema are Collateral status, Clot Burden Score, Vein Score, Change in CSF volume. In this study the specific image findings are manually annotated and also automatically detected using deep learning algorithms. Secondary outcome measures are Sensitivity/Specificity/NPV/PPV of specific imaging findings identified by deep learning algorithms.

CONTACTS AND LOCATIONS:
Overall Officials: Sven Poli, MD MSc, Principal Investigator — sven.poli@uni-tuebingen.de
Locations (19):
- St. John's Hospital, Vienna, Austria
- Germany (17):
  - Charité Universitätsmedizin Berlin, Berlin
  - Universitätsklinikum Bonn, Bonn
  - Fraunhofer- Gesellschaft zur Förderung der angewandten Forschung e.V., Fraunhofer MEVIS, Bremen
  - Universitätsklinikum Düsseldorf, Düsseldorf
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - Klinikum der Medizinischen Hochschule Hannover, Hanover
  - Universitätsklinikum Heidelberg, Heidelberg
  - Universitätsklinikum Leipzig, Leipzig
  - Klinikum der Ludwig-Maximilians-Universität München, Munich
  - Technische Universität München, Munich
  - Universitätsklinikum Münster, Münster
  - Universitätsklinikum Regensburg, Regensburg
  - Klinikum Stuttgart, Stuttgart
  - University Hospital Tuebingen, Tübingen
  - Hertie Institute for AI in Brain Health, Tübingen
  - Universitätsklinikum Ulm, Ulm
  - Universitätsklinikum Würzburg, Würzburg
- BRAINOMIX Limited, Oxford, United Kingdom